CLINICAL TRIAL: NCT05524896
Title: Elucidate Vasodilatory Capacity From Histology-Defined Analysis of Coronary CT Angiography
Acronym: HD-FFRct
Status: Completed | Type: Observational
Sponsor: Elucid Bioimaging Inc. (Industry)
Collaborators: St. Francis Medical Center, New Jersey (Other); The Christ Hospital (Other); Medical University of South Carolina (Other); Mie University (Other)
Responsible Party: Sponsor
Other Study IDs: HD-FFRct
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Low FFR: Invasive FFR value <= 0.8
  Interventions: Device: ElucidVivo
- High FFR: Invasive FFR value > 0.8
  Interventions: Device: ElucidVivo

INTERVENTIONS:
Device: ElucidVivo — Plaque morphology characterization for predicting non-invasive fractional flow reserve (FFR)

SUMMARY:
Coronary CT Angiography (CCTA) may be an ideal modality to fill gaps in understanding the extent and rate of progression coronary artery disease. The investigators have developed an image analysis software ElucidVivo that estimates relevant indices, including fractional flow reserve (FFR) . In this study, the investigators aim to assess the value of ElucidVivo-based plaque morphology characterization for predicting non-invasive FFR in patients with suspected coronary artery disease (CAD) who had undergone clinically indicated coronary CTA and invasive coronary angiography (ICA) for physical FFR measurement.

DETAILED DESCRIPTION:
Invasive FFR is a clinically validated measure of lesion-specific ischemia and is preferred over visual estimation of diameter stenosis for clinical decisions regarding coronary revascularization. FFR derived from coronary CTA (FFRct) using computational fluid dynamics (CFD)-based software has been shown to be a reasonably accurate estimate of invasive FFR and is included in contemporary guidelines as a decision-tool for management of patients with intermediate stenosis on coronary CTA. However, other methods have limitations. It is understood that the burden and type of coronary atherosclerosis, in addition to lumen stenosis, significantly impacts the vasodilatory capacity of the vessel walls which may provide a more interpretable analysis and broader clinical acceptance.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have successfully completed at least one (possibly multiple) CCTA for known or suspected coronary artery disease.
* CCTA was no more than 60 days earlier (and not later)

Exclusion Criteria:

* Subject has a history of percutaneous coronary intervention (PCI) with stent implantation and/or coronary artery bypass grafting (CABG)
* Subject with insufficient CCTA image quality (defined strictly as documented in the ElucidVivo Reading Manual)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects for which a CCTA had been taken within 60 days of invasive coronary angiography with FFR measurements.
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Sensitivity | 1 day
  the ability of a test to correctly identify patients with low FFR
Specificity | 1 day
  the ability of a test to correctly identify people without low FFR

SECONDARY OUTCOMES:
Average Error | 1 day
  Difference of noninvasive result - invasive result

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Buckler, Principal Investigator — Elucid Bioimaging Inc.

IPD SHARING:
Plan to Share IPD: No
We will not share IPD

REFERENCES:
- [Background] Varga-Szemes A, Schoepf UJ, Maurovich-Horvat P, Wang R, Xu L, Dargis DM, Emrich T, Buckler AJ. Coronary plaque assessment of Vasodilative capacity by CT angiography effectively estimates fractional flow reserve. Int J Cardiol. 2021 May 15;331:307-315. doi: 10.1016/j.ijcard.2021.01.040. Epub 2021 Jan 30. PMID 33529657